CLINICAL TRIAL: NCT01181011
Title: A Single-centre, Randomized, Open-label, Three-period Crossover Pharmacokinetic Study of 80 mg Telmisartan / 5 mg Amlodipine Fixed Dose Combination Compared With Its Monocomponents in Healthy Chinese Subjects
Brief Title: Telmisartan, Amlodipine and Combination in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1235.30
Record Dates: First submitted 2010-08-10; First posted 2010-08-13 (Estimated); Results first posted 2012-05-10 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — telmisartan amlodipine combination

ARMS (1):
- amlodipine/telmisartan/combination (Experimental): all patients will be assigned to 6 treatment sequences. cross-over design was adopted to ensure each patient would take amlodipine/telmisartan/combination single dose in randomized order
  Interventions: Drug: amlodipine/telmisartan/combination

INTERVENTIONS:
Drug: amlodipine/telmisartan/combination — patient would take amlodipine(5mg)/telmisartan(80mg)/combination(T80+A5mg) single dose in random order, and each dosage will be separated in 21 days interval.

SUMMARY:
To determine the pharmacokinetic profile of 80 mg telmisartan / 5 mg amlodipine (T80/A5) dose combination after single dose in healthy Chinese subjects.

To determine whether a pharmacokinetic interaction exists between telmisartan and amlodipine, following single doses of 80mg telmisartan (T80), and 5 mg amlodipine (A5) tablet alone and in combination, in healthy Chinese subjects.

To evaluate the safety and tolerability of T80 and A5 alone and in combination in healthy Chinese subjects.

ELIGIBILITY:
Inclusion criteria

1. Healthy males and females
2. Aged between 18 and 45 years
3. Body weight more than 50Kg , and Body Mass Index (BMI ) between 19 and 24 kg/m2

Exclusion criteria

1. Any finding of the medical examination deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker
13. Inability to refrain from smoking during 24 hours prior to dosing and during the trial
14. Alcohol abuse or inability to stop alcoholic beverages for 24 hours prior to dosing and during the trial
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. A history of additional risk factors for torsade de pointes
21. Any history of relevant low blood pressure
22. Supine blood pressure at screening of systolic <110 mm Hg and diastolic < 60 mm Hg
23. History of urticaria
24. History of angioneurotic edema 25 Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion

26. No adequate contraception during the study and until 1 month of study completion 27. Lactation period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1235.30.86001 Boehringer Ingelheim Investigational Site, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 28
Received Telmisartan 80mg | 27
Received Telmisartan 80mg,Amlodipine 5mg | 27
Received Amlodipine 5mg | 26
Completed | 25
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: all patients will be assigned to 6 treatment sequences. cross-over design was adopted to ensure each patient would take amlodipine/telmisartan/combination single dose in randomized order
Arm/Group | All Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Telmisartan in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point (AUC_0-tz)
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for AUC_0-tz of Telmisartan
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 27 | 27
ng·h/mL | 3200 (74.7) | 2940 (94.4)
Statistical Analysis 1: Comparison: Telmisartan 80mg, Amlodipine 5mg vs Telmisartan 80mg; Test type: Non-Inferiority or Equivalence — Bioequivalence; p = 0.0107, ANCOVA — The p-value is for the ratio being outside the interval 0.8 to 1.25; gMean Ratio = 109.22, 90% CI [99.45 to 119.95], Standard Error of Mean 1.06

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From the Time of Dosing to Infinity (AUC_0-∞) of Telmisartan
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for AUC_0-∞ of Telmisartan
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 27 | 27
ng·h/mL | 3420 (82.5) | 3140 (98.5)
Statistical Analysis 1: Comparison: Telmisartan 80mg, Amlodipine 5mg vs Telmisartan 80mg; Test type: Non-Inferiority or Equivalence — Bioequivalence; p = 0.0139, ANCOVA — The p-value is for the ratio being outside the interval 0.8 to 1.25; gMean Ratio = 109.84, 90% CI 2-sided [99.96 to 120.71], Standard Error of Mean 1.06

3. Primary Outcome: The Maximum Observed Plasma Concentration (Cmax) of Telmisartan
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for Cmax of Telmisartan
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 27 | 27
ng/mL | 461 (59.9) | 480 (78.3)
Statistical Analysis 1: Comparison: Telmisartan 80mg, Amlodipine 5mg vs Telmisartan 80mg; Test type: Non-Inferiority or Equivalence — Bioequivalence; p = 0.0126, ANCOVA — The p-value is for the ratio being outside the interval 0.8 to 1.25; gMean Ratio = 97.57, 90% CI 2-sided [84.643 to 112.472], Standard Error of Mean 1.09

4. Primary Outcome: AUC_0-tz of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for AUC_0-tz of Amlodipine
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 27 | 25
ng·h/mL | 206 (28.6) | 192 (31)
Statistical Analysis 1: Comparison: Telmisartan 80mg, Amlodipine 5mg vs Amlodipine 5mg; Test type: Non-Inferiority or Equivalence — Bioequivalence; p = 0.0011, ANCOVA — The p-value is for the ratio being outside the interval 0.8 to 1.25; gMean Ratio = 109.7, 90% CI 2-sided [102.87 to 117.07], Standard Error of Mean 1.04

5. Primary Outcome: AUC_0-∞ of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for AUC_0-∞ of Amlodipine
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 27 | 25
ng·h/mL | 225 (27.1) | 210 (30.9)
Statistical Analysis 1: Comparison: Telmisartan 80mg, Amlodipine 5mg vs Amlodipine 5mg; Test type: Non-Inferiority or Equivalence — Bioequivalence; p = 0.0006, ANCOVA — The p-value is for the ratio being outside the interval 0.8 to 1.25; gMean Ratio = 108.8, 95% CI 2-sided [102.1 to 116.0], Standard Error of Mean 1.04

6. Primary Outcome: Cmax of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days of wash-outs
Population: All patients with values for Cmax of Amlodipine
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 27 | 26
ng/mL | 4.72 (21.7) | 4.43 (27.3)
Statistical Analysis 1: Comparison: Telmisartan 80mg, Amlodipine 5mg vs Amlodipine 5mg; Test type: Non-Inferiority or Equivalence — Bioequivalence; p = 0.000, ANCOVA — The p-value is for the ratio being outside the interval 0.8 to 1.25; gMean Ratio = 106.7, 90% CI 2-sided [100.9 to 112.9], Standard Error of Mean 1.03

7. Secondary Outcome: Time to Attain Cmax (Tmax) of Telmisartan
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for tmax of Telmisartan
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 25 | 25
h | 1.22 (0.58) [0.5 to 3.0] | 1.16 (0.76) [0.5 to 4.02]

8. Secondary Outcome: Terminal Rate Constant in Plasma (λz) of Telmisartan
Description: reflect the speed of drug elimination in vivo
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for λz of Telmisartan
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 25 | 25
1/h | 0.0305 (0.0114) | 0.0323 (0.0124)

9. Secondary Outcome: Mean Residence Time of Telmisartan in the Body After Oral Administration (MRT_po)
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for MRT_po of Telmisartan
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 25 | 25
h | 20.0 (4.8) | 18.4 (5.7)

10. Secondary Outcome: Elimination Half-life (t_½) of Telmisartan
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for t_½ of Telmisartan
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 25 | 25
h | 27.0 (13.7) | 25.0 (10.7)

11. Secondary Outcome: Apparent Clearance of Telmisartan in Plasma Following Extravascular Administration (CL/F)
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for CL/F of Telmisartan
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 25 | 25
L/h | 31.0 (21.6) | 37.3 (39.7)

12. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase λz Following an Extravascular Administration (V_z/F) of Telmisartan
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for V_z/F of Telmisartan
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg
Number analyzed (Participants) | 25 | 25
L | 1021 (697) | 1135 (1018)

13. Secondary Outcome: Tmax of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for tmax of Amlodipine
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 25 | 25
h | 6.88 (1.74) [6.0 to 12.0] | 7.20 (1.63) [6.0 to 12.0]

14. Secondary Outcome: λz of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for λz of Amlodipine
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 25 | 25
1/h | 0.0305 (0.0114) | 0.0323 (0.0124)

15. Secondary Outcome: MRT_po of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for MRT_po of Amlodipine
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 25 | 25
h | 44.3 (7.0) | 43.7 (7.6)

16. Secondary Outcome: t_½ of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for t_½ of Amlodipine
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 25 | 25
h | 38.8 (7.6) | 38.6 (7.5)

17. Secondary Outcome: CL/F of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for CL/F of Amlodipine
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 25 | 25
L/h | 22.7 (6.3) | 25.1 (7.9)

18. Secondary Outcome: V_z/F of Amlodipine
Time Frame: 3 periods of single-dose treatment (8 days of sampling) separated by 21 days wash-outs
Population: All patients with values for V_z/F of Amlodipine
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Amlodipine 5mg
Number analyzed (Participants) | 25 | 25
L | 1241 (313) | 1353 (369)

19. Secondary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event
Time Frame: 4 weeks
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg | Amlodipine 5mg
Number analyzed (Participants) | 27 | 27 | 26
Participants | 4 | 2 | 4

20. Secondary Outcome: Number of Participants With Clinically Relevant Findings in Electrocardiogram (ECG), Vital Signs, Physical Finding or Laboratory Finding Abnormalities
Time Frame: 4 weeks
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg | Amlodipine 5mg
Number analyzed (Participants) | 27 | 27 | 26
Participants
  ECG abnormalities | 0 | 0 | 0
  Vital signs abnormalities | 0 | 0 | 0
  Physical finding abnormalities | 0 | 0 | 0
  Laboratory finding abnormalities | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Telmisartan 80mg, Amlodipine 5mg | Telmisartan 80mg | Amlodipine 5mg
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 2/27 | 1/27 | 3/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 80mg, Amlodipine 5mg (N=27) | Telmisartan 80mg (N=27) | Amlodipine 5mg (N=26)
Influenza (Infections and infestations) | 2 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.